CLINICAL TRIAL: NCT06878495
Title: Optimizing IBD Management: A Comparative Study on the Efficacy and Safety of 5-ASA De-escalation in Patients With Ulcerative Colitis and Crohn's Disease on Stable Biologic or Immunomodulator Therapy
Brief Title: Efficacy and Safety of Discontinuing 5-ASA in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Min Hong, Professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2412-015-145
Record Dates: First submitted 2025-02-02; First posted 2025-03-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis (UC); Crohn's Disease; Inflammatory Bowel Disease (IBD)
Keywords: 5-ASA Discontinuation; Inflammatory Bowel Disease; Biologic Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: 5-ASA Discontinuation Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5-ASA Discontinuation Group (Experimental): The group discontinuing 5-ASA.
  Interventions: Other: Discontinuation of 5-ASA

INTERVENTIONS:
Other: Discontinuation of 5-ASA — Discontinuation of 5-ASA from the time of study enrollment.

SUMMARY:
This study aims to evaluate the long-term outcomes of discontinuing 5-ASA in UC and CD patients receiving stable biologic or immunomodulator therapy using a prospective cohort based in the Busan-Ulsan-Gyeongnam region. It seeks to determine whether discontinuing 5-ASA is a safe treatment strategy in modern IBD management.

DETAILED DESCRIPTION:
In inflammatory bowel disease (IBD), 5-aminosalicylic acid (5-ASA) is widely used as a first-line treatment for ulcerative colitis (UC) and is still prescribed for Crohn's disease (CD). However, for patients who do not respond to conventional therapy, anti-tumor necrosis factor (anti-TNF) agents have become an effective alternative. This has led to ongoing debate about whether continued use of 5-ASA is necessary after transitioning to anti-TNF therapy.

Recent retrospective studies have reported that discontinuing 5-ASA after initiating anti-TNF therapy in UC and CD patients does not increase the risk of clinical adverse outcomes such as new steroid use, hospitalization, or bowel surgery. However, a study based on U.S. data had a median follow-up period of less than one year, making it difficult to assess long-term effects. Additionally, studies on relapse risk after discontinuing 5-ASA have identified younger age, extensive disease, and frequent relapses as risk factors, but detailed analyses for patients receiving anti-TNF therapy remain insufficient.

Another critical issue is the economic burden of continued 5-ASA treatment. In South Korea, the annual cost of the most commonly used 5-ASA formulations constitutes a significant portion of overall healthcare expenses. Discontinuing 5-ASA could reduce treatment costs, simplify therapy, improve patient adherence, and minimize adverse effects associated with polypharmacy. Regarding colorectal cancer (CRC) prevention, recent trends indicate a decreasing incidence of CRC in IBD patients. Since mucosal inflammation is considered a primary driver of CRC, additional 5-ASA use may not be necessary if mucosal healing is achieved through biologics or small-molecule therapies.

Accordingly, this study aims to evaluate the long-term outcomes of discontinuing 5-ASA in UC and CD patients receiving stable biologic or immunomodulator therapy.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis

   o Patients diagnosed with ulcerative colitis (UC) or Crohn's disease (CD) based on standard diagnostic criteria, including clinical, endoscopic, and histologic findings.
2. Treatment Status

   * Patients who have been continuously treated with biologic agents (e.g., anti-TNF agents, integrin inhibitors, JAK inhibitors) or immunomodulators (e.g., azathioprine, methotrexate) for at least three months.
   * Patients who have been on a stable dose of 5-ASA (mesalamine) for at least three months before study enrollment.
3. Disease Activity

   o Patients in clinical remission for at least three months, as defined by the Mayo score for UC or the Crohn's Disease Activity Index (CDAI) for CD.
4. Age

   o Adults aged 19 years or older.
5. Informed Consent

   o Patients capable of providing written informed consent for study participation.
6. Compliance with Study Protocol

   o Patients who can adhere to the study protocol and visit schedule.
7. General Health Condition

   o Patients without severe medical conditions that could impact the study or patient safety, such as significant cardiac, renal, or hepatic diseases.
8. No recent medication changes
9. Patients who have not had any new prescriptions or dose adjustments of corticosteroids, antibiotics, or other medications that could affect IBD within a specified period (e.g., four weeks) before enrollment.

Exclusion Criteria

1. Patients with severe active UC or CD at the time of study enrollment.
2. Patients who have been recently hospitalized for IBD-related reasons or undergone IBD-related surgery within three months before enrollment.
3. Patients who have had dose modifications of biologics, immunomodulators, or corticosteroids for IBD within three months before enrollment.
4. Patients receiving concomitant therapy with other medications that may affect disease activity (e.g., additional anti-inflammatory agents, IBD-related antibiotics).
5. Patients with severe cardiac, renal, or hepatic disease or other medical conditions that could interfere with the study.
6. Pregnant or breastfeeding women.
7. Patients with known allergies or intolerance to 5-ASA or related medications.
8. Patients currently participating in another clinical study that may interfere with this study.
9. Patients unable to provide informed consent or unlikely to comply with the study protocol and visit schedule.
10. Patients with a history of non-response or intolerance to their current biologic or immunomodulator therapy.
11. Patients with a history of severe psychiatric disorders that may affect their ability to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease relapse rate | Through study completion, an average of 9 months

SECONDARY OUTCOMES:
Changes in serum C-reactive protein (CRP) level | Through study completion, an average of 9 months
Changes in fecal calprotectin level | Through study completion, an average of 9 months
Number of hospitalizations | Through study completion, an average of 9 months
Number of emergency department visits | Through study completion, an average of 9 months
Quality of life assessment (32-Item Inflammatory Bowel Disease Questionnaire) | Through study completion, an average of 9 months
  Bowel symptoms (Stool frequency, loose stool, abdominal bloating and pain, excessive flatulence, rectal bleeding, urge to defecate, nausea), Systemic symptoms (Fatigue, lack of energy, sleep problems, weight maintenance, general health), Emotional function (Worry, anxiety, frustration, restlessness, depression, stress, embarrassment, anger), Social function (Ability to engage in social activities, work/school, sexual activity)

CONTACTS AND LOCATIONS:
Overall Officials: Seung Min Hong, M.D., Principal Investigator — Pusan National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seo J, Kim S, Hong SW, Hwang SW, Park SH, Yang DH, Byeon JS, Myung SJ, Yang SK, Kim YJ, Ye BD. Continuing or stopping 5-aminosalicylates in patients with inflammatory bowel disease on anti-TNF therapy: A nationwide population-based study. Aliment Pharmacol Ther. 2024 Aug;60(3):389-400. doi: 10.1111/apt.18102. Epub 2024 Jun 12. PMID 38866064
- [Background] Chapman TP, Frias Gomes C, Louis E, Colombel JF, Satsangi J. Review article: withdrawal of 5-aminosalicylates in inflammatory bowel disease. Aliment Pharmacol Ther. 2020 Jul;52(1):73-84. doi: 10.1111/apt.15771. Epub 2020 May 26. PMID 32452591
- [Background] Singh S, Kim J, Zhu W, Dulai PS, Sandborn WJ, Jairath V. No benefit of continuing vs stopping 5-aminosalicylates in patients with ulcerative colitis escalated to anti-metabolite therapy. Aliment Pharmacol Ther. 2020 Aug;52(3):481-491. doi: 10.1111/apt.15876. Epub 2020 Jun 23. PMID 32573825
- [Background] Ungaro RC, Limketkai BN, Jensen CB, Yzet C, Allin KH, Agrawal M, Ullman T, Burisch J, Jess T, Colombel JF. Stopping Mesalamine Therapy in Patients With Crohn's Disease Starting Biologic Therapy Does Not Increase Risk of Adverse Outcomes. Clin Gastroenterol Hepatol. 2020 May;18(5):1152-1160.e1. doi: 10.1016/j.cgh.2019.08.012. Epub 2019 Aug 13. PMID 31419574
- [Background] Ungaro RC, Limketkai BN, Jensen CB, Allin KH, Agrawal M, Ullman T, Colombel JF, Jess T. Stopping 5-aminosalicylates in patients with ulcerative colitis starting biologic therapy does not increase the risk of adverse clinical outcomes: analysis of two nationwide population-based cohorts. Gut. 2019 Jun;68(6):977-984. doi: 10.1136/gutjnl-2018-317021. Epub 2018 Nov 12. PMID 30420398
- [Background] Bernstein CN, Tenakoon A, Singh H, Targownik LE. Continued 5ASA use after initiation of anti-TNF or immunomodulator confers no benefit in IBD: a population-based study. Aliment Pharmacol Ther. 2021 Sep;54(6):814-832. doi: 10.1111/apt.16518. Epub 2021 Jul 11. PMID 34247410